CLINICAL TRIAL: NCT05410873
Title: Examining the Effects of Mitochondrial Oxidative Stress in DCM
Acronym: MitoDCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21IC6593
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Dilated Cardiomyopathy
Keywords: Energetics; Mitochondria; Oxidative stress
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Experimental): Mitoquinol mesylate 40mg daily
  Interventions: Drug: MitoQ Compound
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MitoQ Compound — Mitoquinol mesylate
  Arms: MitoQ
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Double blind, randomised, placebo-controlled trial of MitoQ (mitoquinol mesylate) in 106 patients with dilated cardiomyopathy, examining the effect of reducing mitochondrial oxidative stress on myocardial energetics and myocardial function using 31-phosphorus magnetic resonance spectroscopy and cardiovascular magnetic resonance.

ELIGIBILITY:
Inclusion criteria

1. idiopathic or familial DCM
2. LVEF ≤45% on 2 imaging studies of any modality ≥3 months apart (may include CMR scan at baseline visit)
3. on guideline therapy for ≥3 months as determined by usual clinicians
4. sinus rhythm on 12-lead electrocardiogram
5. plasma NT-pro-BNP >250ng/L for those >65 years and >100ng/L for those aged ≤65 years within the last 6 months (may include sample at baseline visit)

Exclusion criteria

1. current persistent atrial fibrillation
2. contraindication to CMR
3. estimated glomerular filtration rate (eGFR) <30mls/min
4. current or planned pregnancy or current breast-feeding
5. clear environmental trigger such as excess alcohol intake, cardiotoxic chemotherapy or peripartum presentation
6. fibrosis burden >25% on CMR
7. current cancer (other than non-melanoma skin cancers)
8. current use of CoQ10
9. current participation in another randomised controlled trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Vanguard phase - change in myocardial PCr:ATP | 3 months
  The first 34 patients will enter a 3 months Vanguard phase. Change in myocardial PCr:ATP between baseline and follow-up will be measured using 31P magnetic resonance spectroscopy
Vanguard phase - change in circulating markers of oxidative stress | 3 months
  The first 34 patients will enter a 3 months Vanguard phase. Change in circulating oxLDL and F2isoprostanes will be measured in plasma samples
Primary outcome - change in LVESVi | 12 months
  Change in LVESVi (ml/m2) between baseline and follow-up amongst all 106 patients measured using cardiovascular magnetic resonance

SECONDARY OUTCOMES:
Vanguard phase - change in skeletal muscle PCr recovery | 3 months
  The first 34 patients will enter a 3 months Vanguard phase. Change in skeletal muscle PCr recovery between baseline and follow-up will be measured using 31P magnetic resonance spectroscopy
Follow-on phase - change in LVEF | 12 months
  Change in LVEF (%) between baseline and follow-up amongst all 106 patients measured using cardiovascular magnetic resonance
Follow-on phase - change in LVEDVi | 12 months
  Change in LVEDVi (ml/m2) between baseline and follow-up amongst all 106 patients measured using cardiovascular magnetic resonance
Follow-on phase - change in GLS | 12 months
  Change in GLS between baseline and follow-up amongst all 106 patients measured using cardiovascular magnetic resonance
Follow-on phase - change in NT-pro-BNP | 12 months
  Change in plasma concentrations of NT-pro-BNP (ng/L) between baseline and follow-up amongst all 106 patients
Follow-on phase - change in renal function | 12 months
  Change in creatinine and eGFR between baseline and follow-up amongst all 106 patients
Follow-on phase - change in symptom burden | 12 months
  Change in symptom score between baseline and follow-up amongst all 106 patients
Follow-on phase - change in exercise capacity | 12 months
  Change in 6 minute walk test distance between baseline and follow-up amongst all 106 patients

CONTACTS AND LOCATIONS:
Overall Officials: Brian Halliday, MBChB PhD, Principal Investigator — Imperial College London and Royal Brompton Hospital
Locations (1):
- Royal Brompton Hospital, London, United Kingdom